CLINICAL TRIAL: NCT06816355
Title: Exogenous Sex Hormones and PONV: Evaluating Postoperative Nausea and Vomiting Risk in Transgender Patients
Brief Title: Exogenous Sex Hormones and PONV
Status: Completed | Type: Observational
Sponsor: Riverside University Health System Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Baker, Research Coordinator, Riverside University Health System Medical Center
Other Study IDs: PONV
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Nausea and Vomiting; Sex Hormone; Transgender
Keywords: Postoperative nausea and vomiting; sex hormone; estrogen; testosterone; transgender
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Orchiectomy; Hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Transgender male
  Interventions: Procedure: Hysterectomy
- Transgender female
  Interventions: Procedure: Orchiectomy; Procedure: Augmentation mammoplasty
- Cisgender male
  Interventions: Procedure: Orchiectomy
- Cisgender female
  Interventions: Procedure: Hysterectomy; Procedure: Augmentation mammoplasty

INTERVENTIONS:
Procedure: Orchiectomy — CPT:54520
  Groups: Cisgender male; Transgender female
Procedure: Hysterectomy — CPT:1013911
  Groups: Cisgender female; Transgender male
Procedure: Augmentation mammoplasty — CPT:19325
  Groups: Cisgender female; Transgender female

SUMMARY:
This study aims to investigate the rates of postoperative nausea and vomiting in transgender patients on hormone therapy compared to cisgender patients undergoing the same procedures (hysterectomy, orchiectomy, augmentation mammoplasty).

DETAILED DESCRIPTION:
A retrospective cohort study will be performed using the TriNetX database. Cohorts were defined using Common Procedural Terminology and International Classification of Diseases-10 codes. Separate analyses will be performed for hysterectomies, orchiectomies, and augmentation mammoplasties. Patients will be excluded if they had a history of postoperative nausea and vomiting or a history of neoplasm for which the respective procedure would be indicated (e.g., uterine, cervical, testicular, or breast cancer). Transgender patients will be excluded if not on exogenous hormone therapy and cisgender patients will be excluded if on the same exogenous hormone therapy as their transgender counterparts. Patients will be divided into two groups (transgender group and cisgender group) based on whether they had a diagnosis of sex reassignment, transsexualism, or gender identity disorder. The cohorts will be propensity score-matched based on age, race/ethnicity, and tobacco use.

ELIGIBILITY:
Hysterectomy Cohort:

Inclusion:

- Patients who underwent hysterectomies.

Exclusion:

- Patients who had malignant neoplasm of the uterus, ovarian, cervical, endometrium, or adnexa.

Transgender Male Group

Inclusion:

* administered testosterone within 6 months and 1 day before their hysterectomy
* have one of the following diagnoses: personal history of sex reassignment, gender identity disorders, or transsexualism.

Cisgender Female Group

Inclusion:

- identified as female.

Exclusion:

* administered testosterone within 6 months and 1 day before their hysterectomy
* have one of the following diagnoses: personal history of sex reassignment, gender identity disorders, or transsexualism.

Orchiectomy Cohort:

Inclusion:

- patients underwent an orchiectomy.

Exclusion:

- history of malignant neoplasm of the testis, malignant neoplasm of the prostate, Fournier gangrene, or vascular disorders of male genital organs

Transgender Female Group

Inclusion:

* administered estrogen within 6 months and 1 day before their orchiectomy
* have one of the following diagnoses: personal history of sex reassignment, gender identity disorders, or transsexualism.

Cisgender Male Group

Inclusion:

- identified as male.

Exclusion:

* administered estrogen within 6 months and 1 day before their orchiectomy
* have one of the following diagnoses: personal history of sex reassignment, gender identity disorders, or transsexualism.

Augmentation Mammoplasty:

Inclusion:

- underwent augmentation mammoplasties.

Exclusion:

- Have diagnosis of malignant neoplasm of the breast .

Transgender Female Group

Inclusion:

* administered estrogen within 6 months and 1 day before their augmentation mammoplasty
* have one of the following diagnoses: personal history of sex reassignment, gender identity disorder, or transsexualism.

Cisgender Female Group

Inclusion:

- Identified as female

Exclusion:

* administered estrogen within 6 months and 1 day before their hysterectomy
* have one of the following diagnoses: personal history of sex reassignment, gender identity disorders, or transsexualism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender males, Cisgender females, Transgender males, Transgender females
Study Population: Patients undergoing orchiectomies, hysterectomies, or augmentation mammoplasties.
Sampling Method: Non-Probability Sample
Enrollment: 7348 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Rescue antiemetics | Within 24 hours of surgery
  The primary outcome will be the administration of a rescue antiemetic within 24 hours of surgery. Rescue antiemetics will include droperidol, promethazine, dimenhydrinate, metoclopramide, and prochlorperazine based on rescue antiemetics from the Fourth Consensus PONV Guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Riverside University Health System Medical Center, Moreno Valley, California, United States

IPD SHARING:
Plan to Share IPD: No
A plan to share IPD is not in place at this time.